CLINICAL TRIAL: NCT06325579
Title: Immersive Virtual Reality for Dysphagia Treatment After Stroke
Brief Title: Immersive Virtual Reality for Dysphagia
Acronym: IVRys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: AA29411356
Record Dates: First submitted 2024-02-07; First posted 2024-03-22 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Virtual Reality; Dysphagia; Treatment Compliance
MeSH Terms: conditions — Deglutition Disorders; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dysphagia patients using VR (Experimental): Day 1: Consent taken 5mins. Baseline period wearing strain gauge 5mins, it´d pick up and measure the patient's swallow movements while at rest not using the VR. IVR trial 25mins, the headset will be refitted and instructions to use two different games for up to 10 minutes with a 5-minute break in between. The SALT Assistant would be closely guide and monitor the participant. The experience will be concluded for the day if the participant shows sign of or indicates discomfort.
  Days 2-4 (30-35mins) same proceed as above, minus the test experience (Baseline period (5 mins) and IVR trial (25 mins).
  Day 5 (40-45mins) final day of the trial and after take part in a short semi-structured interview (10mins) in person and audio recorded by the SALT Assistant. SALT Assistant post-trial interview (25-40mins) online audio recorded by a member of the research team .
  Interventions: Device: Immersive Virtual Reality for Dysphagia Treatment

INTERVENTIONS:
Device: Immersive Virtual Reality for Dysphagia Treatment — Patients wore a VR headset while undergoing their rehabilitation session

SUMMARY:
People who have suffered a stroke are at high risk of suffering from oropharyngeal dysphagia with long and intensive exercise programmes. Early access to treatment and engaging therapies is very important for recovery. Immersive virtual reality technology presents an innovative treatment that could help patients improve swallowing. The aim of this study is to improve swallowing in stroke patients using two bespoke immersive virtual reality treatment with real-time feedback. The study consisted in a small feasibility study with stroke patients suffering dysphagia (n = 6, aged of 39 to 80 (M=71.17, SD=15.94). Results obtained through interviews with the patients indicated no discomfort reported during the game. All patients reported enjoying the game and feeling engaged and immersive and four out of six patients reported that they would like to use it every day as part of their Speech and Language therapy. The SALT assistant involved in the study stated that the system had the potential to encourage patients to swallow, being more functional than conventional speech therapy. She identified improvements needed for a better functioning of the VR rehabilitation system for Dysphagia. In a future study, wireless headsets will be used, without a laptop, and it will be important to improve the reliability and design of the strain gauge or innovate in the use of a different technology.

DETAILED DESCRIPTION:
1. Design of the research.

   A priority of the team was to ensure the VR system and game experience is suitable for rehabilitation purposes and use in a clinical setting with OD patients. The research study has been designed collaboratively, with consultations between the research team and relevant clinical staff playing a key role in the development of the IVR intervention. This preliminary work has been further enhanced through:
   * Observation of clinics to establish movements required during rehabilitation.
   * A PPI / expert workshop at early development stage.
   * Play test with healthy volunteers (n = 10) to check usability, acceptability of VR and effectiveness of strain gauge measurement process.
   * Ongoing development informed by consultation with relevant parties and above stages.
2. PPI and contributions. A workshop was conducted which involved people with personal experience of or professional expertise in dysphagia and swallowing problems, which was very valuable in informing and refining the IVR intervention study.

   For this study, further IVR testing sessions were conducted utilising the updated version of the game with healthy adult volunteers. Insights gained from this final stage regarding the enjoyability, usability appropriateness and experience of the scenarios will inform any final amendments to the intervention.
3. Eligibility inclusions and exclusions. The target sample for the clinical feasibility trial was 10 adult (aged 18+) stroke in-patients receiving care at the Stroke.

   Pathway Assessment and Rehabilitation Centre (SPARC) in at STH during the recruitment period of the study.

   In addition to the above, inclusion criteria were comprehension and communication skills sufficient to understand instructions, give informed consent and communicate experiences. Interpreters was provided for people whose first language is not English. People with a mild language or cognitive impairment (common after stroke, which can affect comprehension and communication) was included and supported to participate by the local SALT. People with mild-moderate well-controlled mental health problems could be included, as well as those with a history of mildmoderate motion sickness.

   Exclusion criteria included:
   * A severe language, communication or cognitive impairment preventing full consent or engagement.
   * Hemianopia preventing stereoscopic vision.
   * Severe mental health issues which could give rise to unnecessary, psychological or physical distress during IVR use.
   * Head or neck injuries which would prevent participants wearing the IVR headset and strain gauge around the neck.
   * A history of severe motion sickness since, since IVR can occasionally stimulate motion sickness in those already strongly affected by these symptoms.

   A qualified speech therapist in the SPARC SALT team identified the eligibility of inpatients for the study, based on the above inclusion and exclusion criteria.

   The two members of staff involved in delivering the intervention also took part in interviews following completion of the study.
4. Identification and recruitment of participants. Those who meet eligibility criteria may require information in a more readable, accessible format due to the impact of stroke on some people's ability to comprehend complex information. The full information sheet was designed to be thorough but also clear and easy to read. A second brief information sheet had been developed, in collaboration with a SALT expert, for use with people with mild aphasia, who may find the longer version challenging to follow. This brief version provides the main information about the study and would be reinforced verbally with explanations from a SALT clinician familiar with the full details in the longer comprehensive version of the information sheet.

   Inpatients who were judged to meet the criteria were introduced to the study by a senior SALT or other clinician (e.g.nurse, psychologist) in the SPARC team.

   If the patient expresses interest in hearing more about the study, an information sheet was provided.
5. Informed consent process. There are two versions of the information sheet. The main information sheet provides full details about the study, its inclusion and exclusion criteria, what participation involves and participant rights, including information about withdrawal and confidentiality. It is written to be clear and understandable. A second brief version has been designed and written in an aphasia-friendly way, with support from SALT clinicians, to make it appropriate for people with mild communication or comprehension difficulties. This information sheet was supplemented by verbal explanations from the SALT clinician who provides information, answers questions and takes consent. This clinician was familiar with the comprehensive information in the full information sheet. The full version of the information sheet could also be provided for family / NOK where the brief version had been used with the patient.

   Sufficient time was allowed for the patient to consider the information, ask questions and discuss the study, if they wish, with family members and friends before deciding whether to participate. No pressure was placed upon patients to participate. They were reassured verbally and in the information sheet that deciding against participation would have no consequences whatever for their future treatment.

   Since participation involved the unfamiliar experiences of wearing a VR headset and strain gauge and playing an IVR game, patients who were interested in taking part were offered an opportunity to try out the equipment and experience before making a final decision and giving formal consent.

   After the patient tried out, feels comfortable with the equipment and IVR experience, and wishes to proceed, formal written consent was taken. If the UVR experience or equipment was not comfortable for the patient, they could decide against proceeding, and may indeed be advised not to do so by the SALT Assistant. In this case, they continued with their usual SALT care.

   The SALT staff members involved in the VR trials was invited by email and sent an information sheet about the interview they were asked to attend, with opportunities for questions. Their written consent was taken by email return of a consent form.
6. Right to withdraw. During the recruitment, information-giving and consent-taking process, participants was assured of the right to withdraw from the study at any time, without giving a reason. If participants asked to be withdrawn from the study during or after consent had been taken and procedures started, identifiable data already collected with consent would be retained and used in the study. No further data would be collected, or any other research procedures carried out on or in relation to the participant. This was explained in the information sheet.
7. Risks/burdens and benefits.

   a. Risks:

   - Dizziness and Nausea (a rare side effect of IVR experience in a few people). Some people may find the IVR environment disorientating (e.g. in very early versions there were occasional issues with confusion, nausea, dizziness). To avoid any unnecessary discomfort or distress for participants, it was ensured all those interested in participating had the chance to try out a IVR environment before agreeing to take part. If they felt uncomfortable during the procedure, the IVR could be removed at any stage. They were clearly informed about this before the procedure started and were carefully monitored throughout.

   The SALT assistant worked with the patient each time the IVR is used to ensure that they are comfortable in using the equipment during their SALT session. All practitioners had been trained in using the system prior to the start of the study.

   - Discomfort from the neck band / strain gauge. A specialist company, Footfalls and Heartbeats, had designed a bespoke fabric collar for the purpose of the study, comprising background and sensor yarns. The "background yarn"was composed of interior elastane yarn (6%) and exterior nylon yarn (94%). Both materials were used extensively in clothing. The sensor yarn, a thin gold and black area in the middle of the band, was a plied yarn. This means that two types of yarn were twisted together. None of these yarns were touch the skin of the patient. The yarns were merino wool, the dark colour and a silver (Ag 99.9%) plated polyester yarn, the gold yarn. The band was knitted on a Stoll ADF flatbed knitting machine at Footfalls and Heartbeats (UK) Limited lab in Nottingham. The knitting technique was weft knitting and this allowed for maximum stretch and comfort in the product for the patient.

   Each patient had their own sensor band for the period of the trial. In the unlikely case that washing was required between uses, a careful handwashing process was used. Similar products to these had washed 150 times at 30C in a home environment and the sensor functionality and size and shape of product have continued to function as required.

   Although we couldn't guarantee the band is hypo-allergenic, the Ag coated yarn was unlikely to cause any reaction and was used extensively in medical environments. The nylon base layer fabric was known to create some issues if left on human skin for long periods of time but was routinely used as a medical grade yarn in compression hosiery. Participants would be wearing the band for short periods for the study so allergic reaction is unlikely. The materials used in the band which make skin contact are mentioned in the information sheet.

   As part of the pre-consent checks, participants were offered the opportunity to try out the neck band to see how it feels and decide if it feels comfortable enough to wear during the trial.

   - Infection Control: Each participant had their own dedicated VR kit to use for the duration of their involvement with the trial to prevent cross-infection. In addition, disposable covers was used for the headset, and thorough cleaning took place before and after each use of the equipment. Disinfection took place before and after each set of equipment is allocated to / used by each patient.

   Hospital measures to prevent infection, e.g. from HAIs, Covid-19, were adopted by people involved with the study on all visits to patient, e.g. social distance, PPE, thorough hand washing / sanitisation.

   The VR kit and audio recorder were thorough cleaned and disinfected after use before leaving hospital.

   - Confidentiality of developing software As the study was developing and employing a novel, bespoke intervention, the confidentiality of this product was protected by asking participants to sign non-disclosure agreements at the time of consent. This is explained in the information sheet and explanations was repeated verbally.
8. Confidentiality and anonymity Data collected for the study was treated with the utmost care, stored on password-protected University drives, with non-anonymised and anonymised data files kept separately, with access restricted to the research team.

Hard copy consent forms was kept in locked University cabinets during the study.

Interview audio recordings was deleted from the recorders following their transcription and saved as audio files in password protected computer files, ready for transcription. Some qualitative data extracts were reported verbatim; however personally identifiable details were removed prior to analysis and dissemination; therefore, others should not be able to identify individuals from reports.

It is expected that publications will result from the study; therefore, data will be retained for at least 10 years in the SHU Data Archive (SHURDA) in keeping with the SHU policy on data storage.

ELIGIBILITY:
Inclusion Criteria:

* The target sample for the clinical feasibility trial is 10 adult (aged 18+) stroke in-patients receiving care at the Stroke.

Pathway Assessment and Rehabilitation Centre (SPARC) in at STH during the recruitment period of the study.

In addition to the above, inclusion criteria are comprehension and communication skills sufficient to understand instructions, give informed consent and communicate experiences. Interpreters would be provided for people whose first language is not English. People with a mild language or cognitive impairment (common after stroke, which can affect comprehension and communication) will be included and supported to participate by the local SALT. People with mild-moderate well-controlled mental health problems could be included, as well as those with a history of mildmoderate motion sickness.

Exclusion Criteria:

* A severe language, communication or cognitive impairment preventing full consent or engagement.

  * Hemianopia preventing stereoscopic vision.
  * Severe mental health issues which could give rise to unnecessary. psychological or physical distress during IVR use.
  * Head or neck injuries which would prevent participants wearing the IVR headset and strain gauge around the neck.
  * A history of severe motion sickness since, since IVR can occasionally stimulate motion sickness in those already strongly affected by these symptoms.

A qualified speech therapist in the SPARC SALT team would identify the eligibility of inpatients for the study, based on the above inclusion and exclusion criteria.

The two members of staff involved in delivering the intervention will also take part in interviews following completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the system. Semi-structure Interviews with patients and staffs. Qualitative outcomes. | 10 to 40 minutes interviews
  After the trial to obtain feedback from the patients and speech therapist assistant in the clinical trial, semi structured interviews were use. Questions were focus on their experience of the headset, strain gauge and IVR intervention, and their experiences and perceptions of swallowing whilst playing. Staff questions were focus on her experience of using the IVR with the patient, their perceptions of its effectiveness, usability, potential and limitations.
  Qualitative data was gathered from patient and staff interviews. A qualitative content analysis was conducted to identify the key experiential and perceptual findings.
Feasibility of the system. Semi-structure Interviews with patients. Quantitative outcomes. | 10 to 40 minutes interviews
  The interview will have ten question of liker scales eleven (0-10) answer rate (eg. How comfortable was it to wear the VR headset?; 2. How comfortable was it to wear the strain gauge?).
  Descriptive statistical analyses were conducted using SPSS statistical package.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Phelan, MSc, Principal Investigator — Sheffield Hallam University
Locations (1):
- Sheffield Hallam University, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No